CLINICAL TRIAL: NCT06993064
Title: Effect of Vitamin D Supplementation on Inflammatory Markers in Mexican Population With Type 2 Diabetes Mellitus
Brief Title: Effect of Vitamin D on Inflammatory Markers in Type 2 Diabetes Mellitus in Mexico.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma del Estado de Mexico (Other)
Responsible Party: Principal Investigator, Roxana Valdés Ramos, Doctor in Science, Universidad Autonoma del Estado de Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7236/2025CIB
Record Dates: First submitted 2025-04-29; First posted 2025-05-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes Melitus; Inflammation Biomarkers
Keywords: Type 2 diabetes mellitus; vitamin D supplemention; inflammatory markers
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Longitudinal study of 40 adults with Type 2 Diabetes Mellitus, with six-month follow-up of supplementation with 4000 IU of Vitamin D3/day, with pre and post measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measurement of markers before and after vitamin D supplementation (Other): Measurement of markers before and after vitamin D supplementation
  Interventions: Dietary Supplement: 4000 IU of Vitamin D3

INTERVENTIONS:
Dietary Supplement: 4000 IU of Vitamin D3 — Vitamin D supplementation in Mexican subjects with Type 2 Diabetes Mellitus

SUMMARY:
Type 2 Diabetes Mellitus (T2DM) is a very common disease in Mexico, and its long-term complications affect years of healthy life and a high cost in treatmenty. T2DM is a chronic disease associated to inflammation. We aim to establish if Vitamin D may help decrease this inflammation and improve the condition in adults with T2DM. Patients included in the study will have to take 1 pill/day of vitamin D for six months. The investigators will measure weight, height, waist and hip circumference, systolic and dyastolic blood pressure; obtain dietary and clinical information, as well as a 10mL blood sample from the arm, for laboratory analyses, finger-prick blood sample for glucose at the beginning and end of the study; ´plus a finger-prick blood samplo for the initial vitamin D status. The study is completely free for the participants and they may withdraw their consent at any time without any consequences. Participants will have to attend the clinic at the beginning and every two months until the end, to receive their supplement (total 4 appointments). They will receive a phone call once a week to remind you to take your pills. They will be handed your results at the end of the study.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is the second cause of death in adults of both genders in Mexico, which presents it a as a high public interest pathology. As it is a chronic degenerative disease, it requires long-term treatments and not controlling it leads to the development of important macro and microvascular alterations and ultimately death. There is evidence indicating that the general population all over the world have vitamin D deficiency, which is known to intervene in inflammatory processes associated with most chronic degenerative disease. With respect to T2DM, prolonged low-grade chronic inflammation leads to these associated complications. We hypothesize that 6-month supplementation with 4000 IU/day during 6 months in adults with T2DM will have a positive effect on inflammatory markers, glucose metabolism and lipid profile.

Methods

* Study design Longitudinal study of 40 adults with Type 2 Diabetes Mellitus, with six-month follow-up of supplementation with 4000 IU of Vitamin D3/day, with pre and post measurements.
* Sample

A convenience sample of 40 patients with type 2 diabetes mellitus from community centers in the city of Toluca will be included, according to the following:

Inclusion criteria:

1. Patients medically diagnosed with type 2 diabetes mellitus
2. Patients controlled with diet, metformin or diet and metformin
3. Patients with less than five years of diagnosis
4. Patients with signed informed consent
5. Mexican born from Mexican parents and grandparents
6. Older than 18 years of age.

Elimination criteria:

1. Patients who do not complete the study for any reason
2. Patients that do not comply with the supplementation protocol.

   * Study description

After obtaining approval from the Ethics and Research Committee and authorization from the State of Mexico's Health Institute, subjects from two community health centers will be invited to participate. If compliance with inclusion criteria es fulfilled (18-year-old or more adults with less than five-year medically diagnosed type 2 diabetes, controlled solely with diet, metformin or diet and metformin, Mexican born and being children and grandchildren of Mexican origin), subjects will be asked to sign an informed consent letter. Patients included in the study will be given an appointment for obtaining a finger-prick sample for glucose and a 10mL venous fasting blood sample for biochemical analysis (Insulin, Hb1Ac, Vitamin D, Vitamin D Binding Protein, C-reactive protein, IL-6, total and HDL cholesterol, HOMA-IR will be calculated from insulin and glucose), anthropometric measurements (weight and height for BMI), food-frequency questionnaires, systolic and diastolic blood pressure, as well as general and health information (age, sex, time of diagnosis, treatment, sun-exposure). Subjects will be then given a container with 60 capsules of 4000IU each and given the instructions to consume one daily, they will be given an appointment 60 days later to re-fill the Vitamin D container, this procedure will be repeated on day 120. Every 15 days subjects will receive a reminder phone-call, where compliance will be questioned. After 6 months, the anthropometric, biochemical, dietary and health measurements will be repeated.

After obtaining the blood samples and within one hour of obtention, blood will be centrifuged at 5000 RPM and plasma will be aliquoted into 10 five mL freezer tubes and stored at -70 C for further analysis. Analysis will be done after obtaining all pre- and post-supplementation samples to avoid any differences in the management of samples and to use the same kit for all samples. Insulin, Hb1Ac, Vitamin D, Vitamin D Binding Protein, C-reactive protein, IL-6, total and HDL cholesterol will be analyzed with commercial ELISA-kits.

Results of glucose, blood pressure and anthropometry will be individually given to the study subjects immediately after obtention; results of the intervention measurements will be individually given to patients after finalization of the trial. All data will be maintained confidential, subjects will be given a code number, and all personal information will be kept in a separate database. Any negative effect related to the supplementation will be recorded and reported immediately, in case of danger, supplementation will be suspended, and subject will be referred to their medical doctor.

Statistical analysis Data will be captured into a pre-designed 25.0 SPSS program, after cleaning of the data, we will proceed to analyze the information. Data will be initially described as means, standard deviations, percentiles, frequency or percentages. We will analyze the data with the Shapiro-Wilk test for normality; comparison of initial-final data will be undertaken with paired T-test in the case of parametric data and Wilcoxon for non-parametric data.

ELIGIBILITY:
Inclusion Criteria:

* subjects with medically diagnosed type 2 diabetes mellitus
* controlled with diet and/or metformin
* less than 5 years of evolution
* children and grandchildren of Mexican origin

Exclusion Criteria:

* Subjects that do not complete the study
* Subjects that do not take the supplement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Effect on glycemia | 6 months
  Measurement of glucose at baseline and 6 months
Effect on C-reactive protein | 6 months
  Measurement of C-reactive protein (CRP) before and after supplementation
Effect on glycosilated hemoglobin | 6 months
  Measurement of Hb1Ac at baseline and 6 months
Effect on insulin | 6 months
  Measurement of insulin at baseline and 6 months
Effect on Interleukin 6 | 6 months
  Effect on IL-6 before and after supplementation

SECONDARY OUTCOMES:
Effect on Total Cholesterol | 6 months
  Measurement of Total Cholesterol before and after supplementation
Effect on HDL Cholesterol | 6 months
  Measurement of HDL Cholesterol at baseline and 6 months after supplementation

OTHER OUTCOMES:
Changes on Vitamin D status | 6 months
  Measurement of Vitamin D and Vitamin D binding protein before and after supplementation.
Vitamin D dietary intake | 6 months
  Calculation of Vitamin D dietary intake before and at 6 months after supplementation from food frequency questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Ortíz Reynoso, DPharm, Study Director — Secretary of Research and Graduate Studies. Universidad Autónoma del Estado de México.

IPD SHARING:
Plan to Share IPD: Yes
Age, gender, BMI, body fat, systolic and diastolic blood pressure, vitamin D, vitamin D binding protein, interleukin 6, C-reactive protein, glucose, Hb1Ac, insulin, HDL-cholesterol, total cholesterol, vitamin D intake
Time Frame: Start date: April 2026 End date: April 2028
Access Criteria: The data will be available upon request to the principal investigator.